CLINICAL TRIAL: NCT07300657
Title: Impact of an Artificial Intelligence-Based Chatbot on Implant Patient Management: A Randomised Controlled Trial
Brief Title: Impact of an AI-Based Chatbot on Implant Patient Management: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Marco Cicciù, Full Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Odonto-IA01
Record Dates: First submitted 2025-12-03; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peri-Implant Mucositis; Peri-implantitis; Peri-Implant Health; Peri-implant Inflammation
Keywords: Dental Implants; Oral Hygiene; Artificial Intelligence; Chatbot; Patient Education; Peri-Implant Diseases; Peri-Implantitis; Mucositis; Randomized Controlled Trial; Preventive Dentistry
MeSH Terms: conditions — Peri-Implantitis; Mucositis

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the AI-based chatbot intervention group or the standard oral hygiene education control group. Each participant receives only one intervention during the study. Randomization ensures balanced allocation and reduces selection bias.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Group (Experimental): Participants receive oral hygiene education and motivational support through an AI-based chatbot developed and validated by dental professionals.
  Interventions: Behavioral: AI Chatbot
- Control Group (Active Comparator): Participants receive standard oral hygiene education through printed informational leaflets and scheduled sessions with a dental hygienist.
  Interventions: Behavioral: Standard Oral Hygiene Education

INTERVENTIONS:
Behavioral: AI Chatbot — An artificial intelligence-based chatbot specifically designed and validated by dental experts to provide personalized oral hygiene education and motivational support.
  Arms: Chatbot Group
Behavioral: Standard Oral Hygiene Education — Participants in the Control Group receive traditional oral hygiene education, including printed informational leaflets and scheduled sessions with a dental hygienist.
  Arms: Control Group

SUMMARY:
Background: Dental implant therapy is a well-established and predictable procedure for replacing missing teeth, with high long-term survival rates. However, poor oral hygiene remains one of the main modifiable risk factors for peri-implant diseases such as mucositis and peri-implantitis.

Objective: The aim of this randomized controlled clinical trial is to evaluate the effectiveness of an artificial intelligence (AI)-based chatbot, developed and validated by dental experts, in improving oral hygiene and clinical outcomes in patients with implant-supported restorations, compared to traditional educational methods such as printed leaflets and dental hygienist sessions.

Methods: A total of 110 adult patients rehabilitated with dental implants were randomly assigned to either an AI chatbot intervention group or a control group receiving standard oral hygiene education. The chatbot provides continuous, personalized education and motivation through natural language interaction. Clinical and radiographic parameters, including plaque index (PI), bleeding on probing (BOP), probing pocket depth (PPD), and marginal bone loss (MBL), were recorded at baseline and at follow-up visits.

Expected outcomes: It is hypothesized that the use of an AI-based chatbot will significantly improve oral hygiene compliance and clinical outcomes compared to conventional methods.

Significance: The study aims to demonstrate the potential of AI-assisted patient education in promoting long-term peri-implant health and preventing peri-implant diseases.

DETAILED DESCRIPTION:
Rationale and Background:

Dental implant therapy is highly successful, but peri-implant diseases, primarily caused by inadequate plaque control, remain a major cause of implant failure. Conventional oral hygiene education methods, such as verbal instructions and printed materials, often fail to ensure long-term patient compliance. Artificial intelligence (AI)-based chatbots, powered by large language models, offer a new way to provide continuous, personalized education and motivation to patients. Although their potential has been explored in orthodontics, little is known about their role in peri-implant maintenance.

Study Objective:

This randomized controlled clinical trial investigates whether an AI-based chatbot developed by dental experts can improve oral hygiene compliance and peri-implant health compared to traditional educational methods.

Study Design:

A total of 110 participants were enrolled between June 2024 and June 2025 in private dental practices in Catania, Italy. The study was approved by the local ethics committee (Protocol ID: 60/2024/CL-PAR) and conducted in accordance with the Declaration of Helsinki (2016 revision). Eligible participants were adults (≥18 years), systemically healthy or with controlled conditions, attending regular supportive periodontal therapy, and having at least one osseointegrated implant. Exclusion criteria included active periodontal disease, heavy smoking, systemic immunosuppression, and pregnancy.

Interventions:

Participants were randomly assigned to two groups:

Chatbot group: Received oral hygiene education and motivational support through an AI-based chatbot specifically developed for implant maintenance.

Control group: Received standard oral hygiene instructions through printed materials and sessions with a dental hygienist.

After the study, the chatbot was made available to the control group.

Outcome Measures:

The primary outcome was the Plaque Index (PI) at implant sites. Secondary outcomes included bleeding on probing (BOP), suppuration (SUP), probing pocket depth (PPD), and radiographic marginal bone loss (MBL).

Expected Impact:

This study aims to validate the use of AI-based educational tools as a complementary strategy for improving patient compliance, plaque control, and peri-implant health. The findings could support the safe and effective integration of AI chatbots into clinical dental practice and patient education programs.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy or with controlled systemic conditions;
* Good periodontal health on either an intact or reduced periodontium;
* Regular adherence to supportive periodontal therapy (SPT);
* Presence of at least one osseointegrated dental implant in the maxilla or mandible, following transmucosal healing for 2-4 months;
* Daily access to a smartphone.

Exclusion Criteria:

* Age < 18 years;
* Untreated or active periodontal disease;
* Currently undergoing orthodontic therapy;
* Patients with cognitive deficits;
* Smoking habit (more than 10 cigarettes per day);
* History of heavy alcohol consumption;
* Use of immunosuppressive medication;
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) Score at Implant Sites | Baseline (prosthetic loading of implant) and 6 months after intervention start.
  The PI is considered a direct indicator of the quality of oral hygiene at home and reflects the level of plaque control achieved by each participant. Measurements will be recorded using a standard four-grade scale (0-3) at six sites per implant by a blinded examiner.

SECONDARY OUTCOMES:
Presence of Bleeding on Probing (BOP) at Implant Sites | Baseline (prosthetic loading of implant) and 6 months after intervention start.
  Bleeding on probing (BOP) is used to assess peri-implant tissue inflammation and is defined as the occurrence of bleeding immediately upon probe withdrawal. This parameter will be recorded at six sites per implant.
Presence of Suppuration on Probing (SUP) at Implant Sites | Baseline (prosthetic loading of implant) and 6 months after intervention start.
  Suppuration (SUP) is used to assess peri-implant bacterial infection and is defined as the presence of pus upon probe withdrawal. SUP will be recorded at six sites per implant.
Marginal Bone Loss (MBL) in Millimeters at Implant Sites | Baseline (prosthetic loading of implant) and 6 months after intervention start.
  Marginal bone loss (MBL) will be assessed radiographically at the mesial and distal aspects of each implant and measured in millimeters (mm) to evaluate peri-implant bone level changes over time using standardized periapical radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Intradepartmental Program of Oral Surgery and Early Detection of Oral Cancer, G. Rodolico - San Marco Hospital, AOU Policlinico - San Marco, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including clinical outcomes (Plaque Index, Bleeding on Probing, Probing Pocket Depth) and radiographic outcomes (Marginal Bone Loss), will be shared. Data will be provided in a format suitable for secondary analysis and will exclude any information that could directly identify participants.
Time Frame: IPD and supporting information will be available after publication of the primary study results and will remain accessible for a period of 5 years following publication.
Access Criteria: pubmed